CLINICAL TRIAL: NCT00918112
Title: Development of a Face Valid Executive Functioning Task
Acronym: MedTask
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Parkinson's Disease Association, Inc (Other)
Responsible Party: Sponsor
Other Study IDs: 04-0841
Record Dates: First submitted 2009-06-08; First posted 2009-06-11 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's Disease: Meets criteria for definite Parkinson's Disease
- Healthy Controls: - Must be in good health

SUMMARY:
The purpose of this study is to develop a task to measure executive thinking skills that can be performed in a laboratory setting, but has clear parallels to the thinking demands of real life situations, and can be administered to patients such as those with Parkinson's who have difficulty moving.

ELIGIBILITY:
Brief Inclusion Criteria Parkinson's Disease (PD) group:

* Must have definite PD
* have clear benefit from levodopa

Brief Exclusion Criteria PD Group and Control:

* Hx of stroke
* Head injury
* Visual loss

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruit participants through Volunteer for Health, word of mouth, and from a clinical population at the Washington University in St Louis School of Medicine's Neurological Clinical Research Unit (NCRU).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2004-09; Primary Completion 2009-09 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G Hershey, PhD., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
This was a small pilot study and consent was not obtained to share data.